CLINICAL TRIAL: NCT03978650
Title: Risk Factors for Falls and Fall-related Injuries Associated With Mild Neurocognitive Disorders in the Older Canadian Population: A Population-based, Prospective, Longitudinal, Observational Cohort Study
Brief Title: Risk Factors for Falls and Fall-related Injuries Associated With Mild Neurocognitive Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1804
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Old Age; Fall Injury; Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Participants from the Canadian Longitudinal Study on Aging will be evaluated for cognitive status, occurrence of falls, and fall-related injuries.

SUMMARY:
This study evaluates the risk for incident falls and fall-related injuries at the onset of neurocognitive disorders in older adults participating in the Canadian Longitudinal Study

DETAILED DESCRIPTION:
Falls are frequent events in adults over age 65 (up to 30% each year in Canada). They are a major Canadian public health concern, which negatively impacts health and quality of life of fallers, and health care system. Neurocognitive disorders are strongly associated with falls and fall-related injuries.

Several clinical characteristics, identified previously as risk factors for falls in the older population and in older adults with neurocognitive disorders are selected in the Canadian Longitudinal Study On Aging. The performance criteria of different statistical models will be compared for the association of neurocognitive disorders with falls and fall-related injuries. Six linear statistical models (i.e., logistic regression, discriminant analysis, Bayes network algorithm, decision tree, random forest, boosted trees), Factor Mixture Models and two different artificial neural network (i.e., multilayer perceptron and the neuroevolution of augmenting topologies).

ELIGIBILITY:
Inclusion Criteria:

* People who are 65 years and over
* Men and women who live in Canada

Exclusion Criteria:

* People who do not live in Canada
* A fall resulting from acute medical event and/or an external factor
* Moderate to severe dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: * People from Canada who are 65 years and over.
  * Men and women who were enrolled into the Canadian Longitudinal Study on Aging
  * Participants who attended the face-to-face interview questionnaires about diet, medication use, chronic disease symptoms, and sleep disorders.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Fall Injury | 18 months
  Incident falls occurring during the 18 months. Information related fall- injuries will also be collected, including fractures, dislocations, voluminous intracranial or peripheral hematomas, trauma of the face, and cutaneous lacerations of significant size and/or deeper than the hypodermis, possibly resulting in medical consultation or hospitalization.

SECONDARY OUTCOMES:
Auditory verbal memory disorder | around 20 years
  Investigator will use the Rey Auditory Verbal Test that evaluates the auditory-verbal memory.
The Mental Alteration Test | around 20 years
  Investigator will evaluate the amnesia

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada